CLINICAL TRIAL: NCT05050214
Title: Obinutuzumab for Primary Membranous Nephropathy: a Pilot Study in Patients With Rituximab-resistant or Rituximab-dependent Nephrotic Syndrome and in Patients Intolerant to Rituximab (the ORION Study)
Brief Title: Obinutuzumab in Primary MN
Acronym: ORION
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORION; 2021-004864-81 (EudraCT Number)
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Membranous Nephropathy
Keywords: obinutuzumab; rituximab; membranous nephropathy; B cells; anti-PLA2R
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: GAZYVA, GAZYVARO(Obinutuzumab) (Experimental): Participants will receive Obinutuzumab 1000 mg solution for infusion (total dose of 3000 mg in 30 days).
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — Each patient will be treated for 1 month and received a total of 3 doses. The first dose of Obinutuzumab (1000 mg) will be split in two separate infusions; on the first day each patient will receive 100 mg and the next day 900 mg of Obinutuzumab. Obinutuzumab (1000 mg) will be also administered at two and four weeks after the first infusion. Obinutuzumab will be administered after standard premedication.
  Other Names: GAZYVA; GAZYVARO

SUMMARY:
Primary membranous nephropathy (MN) is an antibody-mediated autoimmune glomerular disease, that represents one of the most frequent causes of nephrotic syndrome in adults. The first-generation chimeric anti-CD20 monoclonal antibody rituximab is effective in inducing MN remission in the majority of patients, but a significant fraction of them can experience disease relapses that require multiple re-treatments over time. Repeated infusions may result in hypersensitivity reactions, which contraindicate further treatment with rituximab. Independent of previous treatment response, Rituximab-Intolerant patients require a safe and effective therapeutic alternative that could reduce the risk of hypersensitivity reactions. On the other end a substantial proportion of patients do not benefit of rituximab therapy and might benefit of other anti CD20 monoclonal antibodies. A few patients transiently benefit of rituximab but their relapses after rituximab administration are so frequent that they spend most of their live with nephrotic range proteinuria (rituximab-dependent patients). Obinutuzumab is a humanized monoclonal antibody with enhanced B cell-depleting potential. Due to humanization and glycoengineering, this drug may be safe and effective in inducing disease remission even in patients with prior hypersensitivity reactions to rituximab. Moreover, it has been found to be effective in patients with membranous nephropathy who failed to respond to rituximab.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years old) on the day of signing informed consent.
2. Biopsy-proven primary membranous nephropathy.
3. Availability of a recent (over the last six months) diagnostic kidney biopsy to confirm the diagnosis of membranous nephropathy and quantify the severity of chronic changes and the number of glomerular podocytes.
4. High-risk of progression to end-stage kidney disease due to persistent nephrotic-range proteinuria (urinary protein excretion > 3.5 g/24-hours as a median of three consecutive measurements) despite background treatment with RAS-inhibitors (ACEi and/or ARBs) at the maximum tolerated doses for at least six months before inclusion.
5. Failure to definitively and effectively respond to rituximab therapy because of the following:

   1. RITUXIMAB-INTOLERANCE, i.e. any previous severe hypersensitivity reaction to rituximab (acute grade III or IV adverse reactions requiring advanced care, or late reactions including delayed serum sickness syndrome) that, independent of response to treatment, preclude further exposure to the drug; or
   2. RITUXIMAB-RESISTANCE: no evidence of nephrotic syndrome complete remission (24-hour proteinuria < 0.3 g/day, normal serum albumin and stable renal function) or partial remission (24-hour proteinuria < 3.5 g/day with > 50% decrease from baseline, normal serum albumin and stable renal function) along with detectable circulating CD19+ lymphocytes for at least 6 months after rituximab administration or
   3. RITUXIMAB-DEPENDENCE: frequently-relapsing nephrotic syndrome (≥ 2 relapses) with nephrotic-range proteinuria for ≥ 50% of time in the 24 months preceding enrolment initial remission after rituximab administration
6. Estimated GFR/eGFR) ≥30 mL/min/1.73 m2 (calculated using the CKD-EPI equation) or qualified endogenous creatinine clearance ≥30 mL/min/1.73 m2 based on 24-hour urine collection during screening.
7. Ability to understand and provide a valid written consent to the study according to the guidelines of the Declaration of Helsinki.
8. Compliance with an effective contraception without interruption, from 28 days before treatment start up to 18 months after treatment discontinuation, agreeing not to donate semen during treatment and for 18 months after discontinuation (if the patient is male), or to undergo pregnancy test during the course of the study (if the patient is female). (According to 2014 CTFG "Recommendations related to contraception and pregnancy testing in clinical trials").

Exclusion criteria:

1. Secondary forms of membranous nephropathy (associated with systemic lupus erythematosus, active hepatitis B, malignancy, drugs such as gold salts and penicillamine, and others).
2. Rituximab treatment or any other prolonged (i.e. for more than two weeks) immunosuppressive treatment in the 6 months preceding anti-CD20 infusion.
3. Uncontrolled hypertension (systolic BP ≥160 and/or diastolic BP >90 mmHg despite therapy).
4. Active bacterial, viral and/or fungal infections.
5. Seropositivity for HIV, regardless of viral load.
6. Active or recent (< 5 years before enrolment) history of malignancy.
7. Known hypersensitivity or allergy to any of the medicaments under investigation.
8. Any other serious medical condition, uncontrolled intercurrent illness or laboratory abnormality that, according to the investigator's judgement, would constitute an unacceptable risk of premature discontinuation from the study.
9. Patients with previous hepatitis B virus infection (seropositive for anti-HBcAb), planning a vaccination with live virus vaccines
10. Known history of drug induced liver injury, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, ongoing extra-hepatic obstruction caused by cholelithiasis, cirrhosis of the liver or portal hypertension.
11. Pregnancy or breast-feeding
12. Childbearing potential and unwillingness or impossibility to comply with a scientifically acceptable birth-control method (According to 2014 CTFG "Recommendations related to contraception and pregnancy testing in clinical trials").
13. Legal incapacity, limited legal capacity, intellectual disability, uncooperative attitude or any other evidence that the patient will not be able to understand the study aims and procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Complete remission or partial remission of nephrotic syndrome. | Changes from baseline and 12 months from Obinutuzumab treatment .
Serious and non-serious adverse events | Through study completion, an average of 24 months.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - ASST HPG23 - Unità di Nefrologia, Bergamo, BG
  - Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica, BG

IPD SHARING:
Plan to Share IPD: No